CLINICAL TRIAL: NCT00341822
Title: Prenatal Testing Decisions in Pregnancy After Infertility
Brief Title: Invasive Prenatal Testing Decisions in Pregnancy After Infertility
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906132; 06-HG-N132
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: Pregnancy
Keywords: Amniocentesis; Chorionic Villus Sampling; Fertility; Genetic Counseling; Decisional Conflict; Prenatal Testing; Questionnaire

SUMMARY:
This study will explore the decision-making experiences of women who are currently pregnant following a period of infertility on whether or not to undergo an invasive prenatal test (IPT) procedure, such as amniocentesis or chorionic villus sampling. Women who become pregnant after infertility often experience heightened anxiety regarding the outcome of the pregnancy. When choosing whether or not to have IPT they are faced with a complex decision, set in the unique context of a pregnancy that they often perceive as exceptionally precarious.

Women who are pregnant with their first child after a period of infertility and have made a decision regarding whether or not to undergo IPT may be eligible for this study.

Participants complete an online password-protected questionnaire that measures infertility and decision-making variables and explores women's perceptions of the impact of infertility on their IPT decision-making process. The questionnaire covers the following areas:

* Subject's demographic information, such as age, marital status, number of children, education, race, ethnicity
* Subject's infertility history
* Subject's thoughts and feelings about infertility
* Subject's thoughts and concerns about other people's (e.g., husband, doctor, other infertile women) opinions about IPT
* Subject's decision about whether or not to have IPT and her feelings regarding the decision
* The effect of subject's infertility history on her decision to have or not have IPT

DETAILED DESCRIPTION:
Women who are pregnant after infertility often experience heightened anxiety regarding the outcome of the pregnancy. When choosing whether or not to have invasive prenatal testing they are faced with a complex decision, set in the unique context of a pregnancy that they often perceive as exceptionally precious. The proposed study aims to explore the invasive prenatal testing decision-making experiences of women who are pregnant after infertility. A cross-sectional design will be used to investigate relationships between the infertility experience and decisional conflict associated with deciding whether or not to have invasive prenatal testing. Women who are pregnant after infertility will be recruited from online support groups and websites for pregnancy after infertility. Participants will be asked to complete a questionnaire that measures infertility and decision-making variables and elicits their perceptions of the impact of infertility on their IPT decision-making experience. The main outcome measure is decisional conflict.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women.

Self-reported history of infertility.

Currently pregnant.

First pregnancy after period of infertility.

Have been offered IPT during current pregnancy for risk of aneuploidy due to maternal age greater than 35 years, abnormal first or second trimester screening or an ultrasound anomaly.

Have made decision about IPT.

Ability to read and write English.

EXCLUSION CRITERIA:

Men, children.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03-29; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Reading AE, Chang LC, Kerin JF. Attitudes and anxiety levels in women conceiving through in vitro fertilization and gamete intrafallopian transfer. Fertil Steril. 1989 Jul;52(1):95-9. doi: 10.1016/s0015-0282(16)60796-3. PMID 2663553